CLINICAL TRIAL: NCT00109512
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of NBI-56418 in Endometriosis
Brief Title: Endometriosis Trial: Study of NBI-56418 in Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-56418-0501
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Endometriosis
Keywords: endometriosis; pelvic pain; painful periods; dysmenorrhea; painful menstruation; GnRH; agonist; antagonist; menstrual pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- NBI-56418 75 mg (Experimental)
  Interventions: Drug: NBI-56418 (GnRH antagonist)
- NBI-56418 150 mg (Experimental)
  Interventions: Drug: NBI-56418 (GnRH antagonist)

INTERVENTIONS:
Drug: NBI-56418 (GnRH antagonist)
  Arms: NBI-56418 150 mg; NBI-56418 75 mg
Drug: placebo
  Arms: placebo

SUMMARY:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled, parallel-group study with subjects randomized to one of three treatment groups, placebo, 75 mg and 150 mg in a 1:1:1 ratio. Study drug was administered once daily for 12 weeks. After the last dose at the end of Week 12, follow-up continued every 4 weeks for 12 weeks.

ELIGIBILITY:
Inclusion Criteria

* Be female, aged 18 to 49 years, inclusive.
* Have pelvic pain and dysmenorrhea resulting in a Composite Pelvic Sign and Symptoms Score (CPSSS) of ≥ 6.
* Have had a diagnosis of endometriosis made following laparoscopic visualization of the disease within the last 5 years of the start of screening.
* Have regular menstrual cycles (28 days ±5 days) for greater than or equal to 2 years. For the cycle that immediately precedes dosing, cycle length will be determined as part of the medical history.
* Have a Body Mass Index between 18 and 30 kg/m2.
* Agree to use two forms of non-hormonal contraception (unless sterilized by tubal ligation) for greater than or equal to 3 months prior to Screening through ovulation and return of menses after treatment.
* Have a negative serum pregnancy test at Screening and a negative urine pregnancy test at prior to dosing at the beginning of Week 1.
* Have a cervical smear negative for malignancy at Screening.
* Be willing to comply with all study procedures and restrictions.
* Be able to read, understand, and sign the ICF (informed consent form) before entering into the study.
* Be willing to provide authorization for access to personal health information in conjunction with US Health Insurance Portability and Accountability Act (HIPAA).

Exclusion Criteria

* Are currently receiving a GnRH agonist or GnRH antagonist, or have received any of these agents within 6 months of Screening.
* Have been nonresponsive to GnRH agonist or antagonist therapy for the management of endometriosis.
* Are currently receiving hormonal therapy including the oral contraceptive pill or have received any of these agents within 3 months of Screening.
* Are on any concurrent medical treatment/medications or have had surgical or hormonal treatment other than oral contraceptives for endometriosis within 3 months of Screening.
* Have uterine fibroids or any other pelvic lesions greater than or equal to 3 cm in diameter as verified by ultrasound.
* Are currently breast-feeding an infant.
* Are using any steroid preparation, taken by any route (e.g., oral, inhaled) on a chronic or regular basis within 3 months of Screening.
* Have an unstable medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary, or endocrine disease), or malignancy that could confound interpretation of the study outcomes.
* Have chronic pelvic pain that is not caused by endometriosis.
* Have any psychological disorder according to criteria indicated in the Diagnostics and Statistical Manual of Mental Disorders, 4th edition within one year before screening. Such disorders include, but are not limited to, alcohol and substance abuse/dependence.
* Have a history of poor compliance in clinical research studies.
* Have a medically significant illness in the 30 days before the beginning of Week 1.
* Have a medically significant abnormality observed upon Screening or the beginning of Week 1 physical examination, or in any other baseline measurement. Findings outside the standard reference ranges will be jointly approved with NBI's (Neurocrine Biosciences) Medical Monitor before being considered eligible for the study.
* Are using any investigational drug within 2 months of Screening.
* Have a positive human immunodeficiency virus antibody (HIV Ab), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCV-Ab) assay at Screening or have a history of a positive result.
* Have an allergy, hypersensitivity, or intolerance to a GnRH agonist or antagonist.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Total Composite Pelvic Signs and Symptom Scale (CPSSS) scores | Every 4 weeks
  This scale is used to assess the signs (pelvic tenderness and induration) and symptoms (nonmenstrual pelvic pain, dysmenorrhea and dyspareunia) associated with endometriosis.

SECONDARY OUTCOMES:
Endometriosis Health Profile-5 (EHP-5) | Every 4 weeks
  The EHP-5 assesses quality of life.
Visual Analog Scale (VAS) scores | Every 4 weeks
  VAS measures endometriosis pain.
Number of Subjects with Adverse Events | Up to 24 weeks
Clinical Laboratory Tests | Up to 24 weeks
Vital Sign Measurements | Up to 24 weeks
Physical Examinations | Up to 24 weeks
Electrocardiogram (ECG) tracings | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura Williams, MD, Study Director — Abbott
Locations (15):
- United States (15):
  - Site Reference ID/Investigator# 56266, Phoenix, Arizona
  - Site Reference ID/Investigator# 55210, San Diego, California
  - Site Reference ID/Investigator# 55214, San Ramon, California
  - Site Reference ID/Investigator# 56267, Clearwater, Florida
  - Site Reference ID/Investigator# 56270, Champaign, Illinois
  - Site Reference ID/Investigator# 56273, Chicago, Illinois
  - Site Reference ID/Investigator# 56269, Oak Brook, Illinois
  - Site Reference ID/Investigator# 56271, Peoria, Illinois
  - Site Reference ID/Investigator# 56272, Louisville, Kentucky
  - Site Reference ID/Investigator# 55213, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 55211, Arlington, Texas
  - Site Reference ID/Investigator# 56268, Sandy City, Utah
  - Site Reference ID/Investigator# 56274, Richmond, Virginia
  - Site Reference ID/Investigator# 55212, Virginia Beach, Virginia
  - Site Reference ID/Investigator# 56275, Spokane, Washington